CLINICAL TRIAL: NCT07264647
Title: Neoadjuvant Chemo-immunotherapy for Stage III PD-L1 Positive Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stage III NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: This is a phase 2 clinical study, monocentric and prospective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- surgery (Experimental): After a neoadjuvant chemoimmuno treatment patient is selected to the surgery and immuno maintenance arm if resectable
  Interventions: Drug: Tislelizumab; Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- chemoradio (Active Comparator): After neoadjuvant chemoimmuno treatment patient is selected to surgery and immuno maintenance arm if resectable
  Interventions: Drug: Tislelizumab; Radiation: Chemoradiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Compared to clinical practice in Italy this trial is adding a neoadjuvant chemoimmuno treatment with adjuvant immuno
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — surgery if resectable after neoadjuvant treatment
  Arms: surgery
Radiation: Chemoradiotherapy — if patient not resectable after neoadjuvant treatment, chemoradiotherapy performed
  Arms: chemoradio

SUMMARY:
A Ph.2, single-arm, monocentric, trial of neo-adjiuvant chemo-immunotherapy for stage III, PD-L1 positive, NSCLC.

Adults and smokers (past or current) diagnosed with stage III NSCLC without driver molecular alterations (EGFR, ALK, ROS1, RET).

DETAILED DESCRIPTION:
Study Population: Adult smoker (past or current) patients diagnosed with stage III (NON T4 for a nodule in a different lobe) NSCLC without driver molecular alterations (EGFR, ALK, ROS1).

Treatment: Patients will receive neoadjuvant chemo-immunotherapy based on NSCLC histology.

Diagnostic Assessments: All patients will undergo a comprehensive disease staging, including contrast-enhanced chest CT, PET-CT, and contrast-enhanced brain magnetic resonance imaging. A pathological assessment of the mediastinum and lymph-node stations clinically positive/suspected is mandatory.

Treatment Cycles: Eligible patients will receive 3 cycles of neoadjuvant chemo- immunotherapy, followed by a comprehensive diagnostic assessment using chest CT and PET-CT and pathologic lymph-node reassessment.

Intervention: Patients with pathologic negativization of lymph nodes after neoadjuvant therapy will be candidate for surgery. Patients with pathologic persistence of N2 or N3 disease will be candidate for definitive concurrent chemoradiation as part of routine clinical practice. After local therapy, patients will receive 1 year of adjuvant or maintenance tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III disease.

  * PD-L1 TPS ≥ 1% according to local testing.
  * No evidence of EGFR mutations or ALK or ROS1 or RET rearrangements by local testing.

Mandatory baseline multidisciplinary assessment to confirm suitability of patient to local treatment with curative intent.

* Pulmonary function tests within 6 months of the planned resection.
* At least 1 measurable lesion as defined by RECIST v1.1.
* ECOG Performance Status ≤ 1.
* Eligibility to receive a platinum doublet chemotherapy regimen.
* Adequate organ function as indicated by the following laboratory values obtained ≤ 14 days before the first dose of study drug:

Patients must not have required blood transfusion or growth factor support ≤ 14 days before sample collection at screening for the following:

Absolute neutrophil count ≥ 1.5 x 109 /L Platelets ≥ 75 x 109 /L Hemoglobin ≥ 90 g/L Estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation (Appendix 9).

For patients intended to receive cisplatin: creatinine clearance 60mL/min For patients intended to receive carboplatin: creatinine clearance 45mL/min Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome).

AST and ALT ≤ 2.5 x ULN For patients not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time 1.5ULN

* Age ≥ 18 years.
* Written informed consent.

Exclusion Criteria:

Evidence of stage IV NSCLC (metastatic disease).

* Histology of large cell neuroendocrine carcinoma (LCNEC).
* Any previous therapy for current lung cancer, including chemotherapy or radiation therapy.
* Previous treatment with an antibody or drug against the immune checkpoint pathway, including but not limited to, therapeutic anti-cytotoxic T-lymphocyte antigen-4-associated antibodies (anti-CTLA-4), anti-PD-1 and anti-PD-L1.
* Never smoking patients.
* Active autoimmune diseases or history of autoimmune diseases that may recur.
* Concomitant participation in another therapeutic clinical trial.
* Pregnancy or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
radical surgery (R0) in patients with stage III PD-L1 positive | 3 years
  To evaluate the rate of radical surgery (R0) in patients with stage III PD-L1 positive NSCLC treated with tislelizumab plus platinum-based doublet chemotherapy as neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cappuzzo, Principal Investigator — Istituti Fisioterapici Ospitalieri
Locations (1):
- Istituti Fisioterapici Ospitalieri, Rome, Roma (RM), Italy